CLINICAL TRIAL: NCT04146818
Title: Study of the Effects of Adapted Tango and Multidimensional Intervention in pREvention of Dementia in agiNG: Developing healTHy Life Style Programs. (STRENGTH)
Brief Title: Study of the Effects of Adapted Tango and Multidimensional Intervention in pREvention of Dementia in agiNG (STRENGTH)
Acronym: STRENGTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INRCA_04_2019; GR-2016-02363041 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; adapted Tango dancing; elderly people; music therapy; psycho-education
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Tango Dancing arm (Experimental): Treatment will include sessions of Adapted Tango (90 min per week for a total of 6 months) together with sessions of comprehensive cognitive intervention (90 min per week for a total of 6 months)
  Interventions: Behavioral: Adapted Tango Dancing
- Control arm (Placebo Comparator): Sessions of psycho-education and advice on healthy life-style (once per month for a total of 6 months)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Adapted Tango Dancing — Treatment will include sessions of Adapted Tango (90 min per week for a total of 6 months) together with sessions of comprehensive cognitive intervention (90 min per week for a total of 6 months) consisting in music therapy, engagement in social activities, cognitive training and psycho-education.
  Arms: Adapted Tango Dancing arm
Behavioral: Control — Sessions of psycho-education and advice on healthy life-style (once per month for a total of 6 months)
  Arms: Control arm

SUMMARY:
The STRENGTH project is a randomized controlled trial to assess the effects of a 6 months multimodal intervention consisted of adapted Tango dancing together with music therapy, engagement in social activities, cognitive intervention and psycho-education on functional, biological, cognitive outcomes and psycho-social aspects in 300 subjects with mild cognitive impairment.

DETAILED DESCRIPTION:
Cognitive decline represents a pathological condition for elderly with negative consequences on social functioning and independent living. To reduce the incidence of cognitive deficits in mild cognitive impairment (MCI), treatments that prevent or delay dementia are needed. The main objective of STRENGTH Project, is the assessment of the effects of a comprehensive intervention in 300 subjects with MCI, finalized to improve functional, biochemical, cognitive outcomes and psycho-social aspects. The study uses a multidisciplinary approach, has a 3-year duration, and includes 3 follow-up phases. Participants will be assigned to: a) Experimental group, which will undergo a multimodal intervention for improving cognitive outcomes, functional status and mobility. Treatment will include sessions of Adapted tango, music therapy, engagement in social activities, comprehensive cognitive intervention and psycho-education for 6 months; or b) Control group, which will receive psycho-education and advice on healthy life-style for 6 months. Cognitive and psycho-social outcomes, functional, cardiovascular status, life-style characteristics, biochemical determination, will be evaluated at baseline and longitudinally. Our hypothesis is based on expectation that the proposed could improve cognitive, functional outcomes and quality of life, with a positive impact on prevention of onset of dementia and cognitive decline in MCI subjects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild cognitive impairment
* presence of a caregiver
* capability to sign the informed consent

Exclusion Criteria:

* diagnosis of dementia
* serious medical and/or psychiatric conditions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2024-06-29 (Estimated); Study Completion 2024-06-29 (Estimated)

PRIMARY OUTCOMES:
change in overall cognition | baseline, 6 months, 12 months and 24 months
  Italian version of the Corsi test. This is a neuropsychological instrument, for the assessment of the spatial learning and memory processes. It consists of 9 blocks randomly arranged on a board. The investigator points to a series of blocks at a rate of one block per second, and then the subjects have to point at the same blocks in the same order. The longest sequence correctly reproduced represents the measure of spatial span. An increase of at least 1 point will indicate the success of the intervention.

SECONDARY OUTCOMES:
change in cognitive status | baseline, 6 months, 12 months and 24 months
  Italian version of the Mini Mental State Examination (MMSE)
change in level of cognitive impairment | baseline, 6 months, 12 months and 24 months
  Clinical Dementia Rating Scale (CDR). An overall Global CDR® Score may be calculated through the use of an CDR® Scoring Algorithm. This score is useful for characterizing and tracking a patient's level of impairment/dementia: 0 = Normal; 0.5 = Very Mild Dementia; 1 = Mild Dementia; 2 = Moderate Dementia; 3 = Severe Dementia.
change in depressive symptoms | baseline, 6 months, 12 months and 24 months
  Geriatric depression scale (GDS-15 items). The score ranges from 0 to 15 and a score of zero to four is considered to be within the normal range, five to nine indicates mild depression, and a score of 10 or more indicates moderate to severe depression.
change in functional status | baseline, 6 months, 12 months and 24 months
  Basic Activities of daily living (BADL). There are 6 domains of function measured with the BADL scale. A summary score ranges from 0 (low function, dependent) to 6 (high function, independent).
change in functional performance | baseline, 6 months, 12 months and 24 months
  Instrumental Activities of Daily Living (IADL). There are 8 domains of function measured with the Lawton IADL scale. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent).
change in social supports | baseline, 6 months, 12 months and 24 months
  Lubben Social Network Scale (LSNS). From the sum of the scores of the 11 items derive four categories: 0-19 poor social support (social isolation); 20-25 discreet support; 26-39 good support; > 40 excellent support.
change in the physical performance | baseline, 6 months, 12 months and 24 months
  6 Minute Walk Test (6MWT). The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
change in psychological well being | baseline, 6 months, 12 months and 24 months
  Psychological well being scales (PWB). PWB is a 84 item self-rating inventory, which consists of six scales which represent the six dimensions of psychological well-being: self-acceptance, autonomy, environmental mastery, personal growth, purpose in life and positive relations.Respondents rate how strongly they agree or disagree with the statements using a 6-point scale (1 = strongly agree; 6 = strongly disagree).
change in quality of life | baseline, 6 months, 12 months and 24 months
  36 Health Survey
change in genetic biomarkers | baseline, 6 months, 12 months and 24 months
  assessment of cellular (leukocytes) microRNA of genes involved in the neurodegeneration process
change in trace elements | baseline, 6 months, 12 months and 24 months
  Identification of trace elements (Zn, Cu, Fe, Se) by flame atomic absorption spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Giuli, PhD, Principal Investigator — IRCCS INRCA
Locations (1):
- Cinzia Giuli, Fermo, Italy

IPD SHARING:
Plan to Share IPD: No